CLINICAL TRIAL: NCT05425719
Title: A Pivotal, Open Label, Multi-Center, Safety and Pharmacokinetic Study of MB-102 (Relmapirazin) and the Use of the MediBeacon Transdermal GFR Measurement System in Normal and Renal Compromised Subjects for the Evaluation of Kidney Function
Brief Title: Pharmacokinetics and Safety of MB-102 (Relmapirazin) and the MediBeacon Transdermal GFR Measurement System in Evaluation of Kidney Function in Normal and Renal Compromised Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MediBeacon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MB-100-003
Record Dates: First submitted 2022-04-21; First posted 2022-06-21 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Disease
Keywords: Glomerular Filtration Rate; Transdermal fluorescence detection; Relmapirazin
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — relmapirazin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- eGFR ≥ 70 mL/min/1.73 m^2 (Experimental): Participants with eGFR ≥ 70 mL/min/1.73 m^2 received one 130 mg dose of MB-102 and a transdermal sensor was placed on their chest. Blood samples and fluorescent measurements were collected over 12 hours.
  Interventions: Drug: MB-102; Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (TGFR)
- eGFR < 70 mL/min/1.73 m^2 (Experimental): Participants with eGFR < 70 mL/min/1.73 m^2 received one 130 mg dose of MB-102 and a transdermal sensor was placed on their chest. Blood samples and fluorescent measurements were collected over 24 hours.
  Interventions: Drug: MB-102; Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (TGFR)

INTERVENTIONS:
Drug: MB-102 — 18.6 mg/mL in a 7.0 mL volume administered by intravenous injection over 30 - 60 seconds, followed by a 10 mL normal saline flush administered intravenously over 30 - 60 seconds
  Other Names: Relmapirazin
Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (TGFR) — On treatment day, participants had a transdermal sensor placed on their upper chest, and the MediBeacon Transdermal GFR Measurement System was initiated to collect background fluorescence. After collection of background fluorescence, participants received a single dose of MB-102.

SUMMARY:
The goal of this clinical trial was to compare transdermal glomerular filtration rate (tGFR) to plasma-derived indexed (to body surface area; BSA) GFR (nGFR) using MB-102 (relmapirazin) as the fluorescent compound. Adults with kidney function ranging from normal to Stage 4 chronic kidney disease (CKD) and participants spanning the entire range of human skin colors as defined by the Fitzpatrick Skin Scale (FSS) were included in the study.

The main questions that the study aimed to answer were:

* To establish that the MB-102 transdermal fluorescence measured GFR using the MediBeacon Transdermal GFR Measurement System is comparable to the measured MB-102 plasma GFR
* To evaluate the safety and tolerability of a single dose of MB-102 in study participants
* To evaluate the safety and effectiveness of the MediBeacon Transdermal GFR Measurement System (TGFR) for the non-invasive transdermal fluorescence detection of MB-102 in participants

Participants had a transdermal sensor placed on their upper chest, and the TGFR collected background fluorescence. Participants then received a single dose of MB-102. Blood samples were collected and fluorescent measurements were taken over a 12- to 24-hour period. Following completion of the treatment period, participants returned to the study center approximately 1 week later for a safety follow-up visit. Researchers compared the results to see if the transdermal GFR measurements were comparable to the measured plasma GFR in those with and without normal kidney function and different skin coloration.

ELIGIBILITY:
Inclusion Criteria:

* Eligible female non-pregnant participants who are either not of child-bearing potential or willing to use adequate contraception during the trial
* Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 7 days post-dose
* For women of child-bearing potential, the participant should have a negative serum pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly i.e. abstinence, oral contraceptive either combined or progesterone alone; injectable progesterone, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, IUD device or system or male partner sterilization
* Men will not donate sperm during the study and for 1 month following the last dose of study drug
* Participants who are capable of directly providing informed consent and who can comply with the requirements and restrictions required by the protocol
* Adequate venous access sufficient to allow blood sampling per protocol requirements

Exclusion Criteria:

* Participants positive via PCR testing for COVID-19 (Vaccinated participants without symptoms of COVID-19 are not required to undergo PCR testing but may be tested at the discretion of the study site)
* Recent donation or loss of blood or plasma: 100 mL to 499 mL within 30 days prior to the initial dose of the study medication; or more than 499 mL within 56 days prior to the initial dose of study medication
* Non-steroidal anti-inflammatory (NSAID) use within 3 days of MB-102 dosing
* Participant has participated in a clinical trial and has received an investigational product within the following time ranges: prior to the first dosing day in the current study: either 30 days or 5 half-lives of the investigational product (whichever duration is longer)
* History of skin sensitivity to adhesives (e.g. Band-Aids, surgical tape)
* History of severe allergic hypersensitivity reactions (unacceptable adverse events) or anaphylactoid reaction to any allergen including drugs, MB-102 or other related products (intolerance to a drug is not considered a drug allergy).
* Any characteristics which, in the opinion of the investigator, makes the participant a poor candidate for participation in the clinical trial
* Significant scarring, tattoos or alterations in pigmentation on the sternum or other sensor location testing areas that would alter sensor readings versus other areas of the skin
* Any serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, or psychiatric condition that in the opinion of the investigator would limit the participant's ability to complete study requirements or may put the participant at increased risk or compromise the interpretability of study results.
* Currently receiving dialysis
* Currently anuric
* Positive serum pregnancy test
* Participants with an eGFR > 120 mL/min/1.73m^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Dorshow, PhD, Study Director — MediBeacon, Inc.
Locations (8):
- United States (5):
  - Velocity Clinical Research, Edgewater, Florida
  - Research by Design, LLC, Chicago, Illinois
  - Nucleus Network, Saint Paul, Minnesota
  - Carolina Phase I Research, Raleigh, North Carolina
  - Endeavor Clinical Trials, LLC, San Antonio, Texas
- China (3):
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Peking University First Hospital, Beijing
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan G, Pino CJ, Johnston KA, Humes HD. Estimating Changes in Glomerular Filtration Rate With Fluorescein Isothiocyanate-Sinistrin During Renal Replacement Therapy. ASAIO J. 2023 Aug 1;69(8):810-815. doi: 10.1097/MAT.0000000000001947. Epub 2023 Apr 27. PMID 37104481

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety Population: all participants who enrolled in the study and were dosed with MB-102
Period: Overall Study
Arm/Group | eGFR ≥ 70 mL/Min/1.73 m^2 | eGFR < 70 mL/Min/1.73 m^2
Started | 130 | 119
Completed | 125 | 118
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrew consent | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: all subjects who enrolled in the study and were dosed with MB-102
Groups:
- Total: Total of all reporting groups
Arm/Group | eGFR ≥ 70 mL/Min/1.73 m^2 | eGFR < 70 mL/Min/1.73 m^2 | Total
Number analyzed (Participants) | 130 | 119 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (14.19) | 61.5 (13.45) | 53.9 (15.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 45 | 107
  Male | 68 | 74 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 14 | 50
  Not Hispanic or Latino | 94 | 103 | 197
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 37 | 27 | 64
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 43 | 76
  White | 58 | 49 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Transdermal Derived Glomerular Filtration Rate (tGFR) Values Within 30% of the nGFR Plasma-derived Indexed Glomerular Filtration Rate (nGFR) Values
Description: The performance measure of P30 is defined as the proportion of transdermal derived GFR values that are within 30% of the measured plasma-derived GFR. The comparison of transdermal derived glomerular filtration rate (tGFR) with respect to the plasma-derived indexed glomerular filtration rate (nGFR) was calculated with a double-sided 95% confidence interval (CI). The performance goal was 0.85, and success for the study was defined as a lower limit of the 95% CI greater than 0.85.
Time Frame: Up to 24 hours following the study dose
Population: Modified intent-to-treat population (all participants enrolled in the study for whom an average session tGFR had been calculated, with no major protocol deviations and no outlier pharmacokinetic parameters)
Measure: Number (95% Confidence Interval); unit: Proportion of tGFR within 30% of nGFR
Groups:
- All Participants: Participants received one 130 mg dose of MB-102 and a transdermal sensor was placed on their chest. Blood samples and fluorescent measurements were collected over 12 - 24 hours.
Arm/Group | eGFR ≥ 70 mL/Min/1.73 m^2 | eGFR < 70 mL/Min/1.73 m^2 | All Participants
Number analyzed (Participants) | 90 | 92 | 182
Proportion of tGFR within 30% of nGFR | 0.96 [0.89 to 0.99] | 0.92 [0.85 to 0.97] | 0.94 [0.89 to 0.97]

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Associated With MB-102 Administration
Description: An adverse event is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, temporally associated with the use of a medicinal product, whether or not related to the investigational medical device or drug.
Time Frame: From the time of dosing through the follow-up visit, up to 10 days
Population: Safety Population: all participants who enrolled in the study and were dosed with MB-102
Measure: Count of Participants; unit: Participants
Arm/Group | eGFR ≥ 70 mL/Min/1.73 m^2 | eGFR < 70 mL/Min/1.73 m^2
Number analyzed (Participants) | 130 | 119
Participants | 1 | 0

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Associated With the MediBeacon Transdermal GFR Measurement System Device
Description: as for outcome 2
Time Frame: From the time of dosing through the follow-up visit, up to 10 days
Population: Safety Population: all participants who enrolled in the study and were dosed with MB-102
Measure: Count of Participants; unit: Participants
Arm/Group | eGFR ≥ 70 mL/Min/1.73 m^2 | eGFR < 70 mL/Min/1.73 m^2
Number analyzed (Participants) | 130 | 119
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the time of dosing through the follow-up visit, up to 10 days
Arm/Group | eGFR ≥ 70 mL/Min/1.73 m^2 | eGFR < 70 mL/Min/1.73 m^2
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/119
Other Adverse Events (participants affected / at risk) | 3/130 | 7/119
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | eGFR ≥ 70 mL/Min/1.73 m^2 (N=130) | eGFR < 70 mL/Min/1.73 m^2 (N=119)
Cardiac murmur (Investigations) | 0 | 2
Headache (Nervous system disorders) | 3 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MediBeacon requests that no presentation/publication occur until after the first publication of study results or until 1 yr after a study is completed/terminated early, whichever occurs first. Proposed results publication/disclosure must be given to Sponsor for review at least 45 days prior to the date of submission. If a patent application is to be filed, both the Institution and the Sponsor will defer publication or other disclosure for a period of time, not to exceed an additional 60 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT05425719/Prot_SAP_001.pdf